CLINICAL TRIAL: NCT03062462
Title: Half-dose Ticagrelor Overcomes High-dose Clopidogrel in Acute Coronary Syndrome Patients With High On-Clopidogrel Platelet Reactivity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCAD-20170220
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease; Clopidogrel, Poor Metabolism of
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- clopidogrel (Active Comparator): To observe double standard-dose clopidogrel on platelet aggregation in clopidogrel resistance's patients with coronary heart disease
  Interventions: Drug: Clopidogrel
- ticagrelor (Experimental): To observe low-dose of ticagrelor on platelet aggregation in clopidogrel resistance's patients with coronary heart disease
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — double standard-dose clopidogrel treatment (300 mg loading dose, then 75 mg twice daily) for 5-7 days
  Arms: clopidogrel
Drug: ticagrelor — half-dose ticagrelor treatment (90 mg loading dose, then 45 mg twice daily) for 5-7 days
  Arms: ticagrelor

SUMMARY:
With the widespread use of clopidogrel, resistance to clopidogrel has been attracting increasing attention, and emerged as a new challenge adversely affecting patients clinical risk and outcome. Clopidogrel resistance means that blood platelets show little or no response to clopidogrel. It is closely associated with increased risk of serious cardiovascular events, seriously affects the prognosis of patients, and brings difficulties to clinical treatment.

Guideline recommendations on the use of dual antiplatelet therapy have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for ACS patients. Recent study found that ticagrelor 90mg twice a day orally could significantly reduce the occurrence of clopidogrel resistance and adverse cardiovascular events. The previous studies have reported that half-dose ticagrelor had the similar inhibitory effect on platelet aggregation as the standard-dose ticagrelor, which was significantly stronger than that in the clopidogrel group. But it is still not very clear that the effect of low-dose ticagrelor on platelet function in patients with clopidogrel resistance and coronary heart disease.

Therefore, we performed this randomized, single-blind clinical trial to observe the effects of low-dose ticagrelor and double standard-dose clopidogrel on platelet aggregation and prognosis in clopidogrel resistance's patients with coronary heart disease.

DETAILED DESCRIPTION:
Dual Antiplatelet Therapy (DAPT) with aspirin and P2Y12 receptor inhibitor remains a cornerstone in the secondary prevention of coronary artery disease (CAD). Clopidogrel is one of the most commonly used antithrombotic agent that inhibits the platelet P2Y(12) adenosine diphosphate (ADP) receptor. With the widespread use of clopidogrel, resistance to clopidogrel has been attracting increasing attention, and emerged as a new challenge adversely affecting patients clinical risk and outcome. Clopidogrel resistance means that blood platelets show little or no response to clopidogrel. Recent studies have found that clopidogrel resistance rate was about 11% ~ 44%. Clopidogrel resistance is more common in patients with loss-of-function CYP2C19 genotypes, and closely associated with increased risk of serious cardiovascular events, including ischemic events, myocardial infarction, stent thrombosis, revascularization and so on. This seriously affects the prognosis of patients, and brings difficulties to clinical treatment.

Ticagrelor is an oral, reversibly-binding, direct-acting P2Y12 receptor antagonist used clinically for the prevention of atherothrombotic events in patients with acute coronary syndromes (ACS). Guideline recommendations on the use of dual antiplatelet therapy have been formulated that ticagrelor 90 mg twice daily plus aspirin in preference to clopidogrel 75mg daily plus aspirin for ACS patients. Recent study found that ticagrelor 90mg twice a day orally could significantly reduce the occurrence of clopidogrel resistance and adverse cardiovascular events. The previous studies have reported that half-dose ticagrelor had the similar inhibitory effect on platelet aggregation as the standard-dose ticagrelor, which was significantly stronger than that in the clopidogrel group. But it is still not very clear that the effect of low-dose ticagrelor on platelet function in patients with clopidogrel resistance and coronary heart disease.

Therefore, we performed this randomized, single-blind clinical trial to observe the effects of low-dose ticagrelor and double standard-dose clopidogrel on platelet aggregation and cardiovascular prognosis in clopidogrel resistance's patients with coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with oral clopidogrel treatment admitted to hospital within 24 hours or long-term follow-up outpatients with oral clopidogrel treatment;
2. The platelet aggregation rate (PAgR) measured with light transmission aggregometry (LTA) is decreased no more than 10% from baseline level, or PAgR is more than 46% and the percentage of inhibition of ADP-induced platelet aggregation measured by thrombelastogram is not more than 30%;

Exclusion Criteria:

1. Planned use of glycoprotein IIb/IIIa receptor inhibitors, adenosine diphosphate (ADP) receptor antagonists, or anticoagulant therapy during the study period;
2. Platelet count <100g/L;
3. Creatinine clearance rate < 30ml/min;
4. Diagnosed as respiratory or circulatory instability (cardiac shock, severe congestive heart failure NYHA II-IV or left ventricular ejection fraction < 40%);
5. A history of bleeding tendency;
6. Aspirin, ticagrelor or clopidogrel allergies;
7. Severe liver injury.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The platelet aggregation rate | up to 7 days
  Light transmission aggregometry method

SECONDARY OUTCOMES:
Side effects including bleeding,dyspnea and arrhythmia | up to 7 days, 1 month, 3 months, 6 months and 12 months
Adverse events including myocardial infarction, death, stroke, re-hospitalization for cardiovascular diseases and ischemia events | up to 7 days, 1 month, 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- whole blood lumi-aggregometer type 560 VS, Havertown, Pennsylvania, United States

REFERENCES:
- [Derived] Liu GZ, Zhang S, Sun DH, Shi J, Bo WL, Wang WN, Zhang CY, Wang ZH, Feng W, He MJ, Liu YY, Li S, Zheng LQ, Li Y. Half-dose ticagrelor versus high-dose clopidogrel in reducing platelet reactivity in acute coronary syndrome patients with high on-clopidogrel platelet reactivity (divide study). Eur J Clin Pharmacol. 2019 Aug;75(8):1059-1068. doi: 10.1007/s00228-019-02687-0. Epub 2019 May 12. PMID 31081522